CLINICAL TRIAL: NCT02287532
Title: Evaluation of the DIABEO System in Poorly Controlled DM1 or DM2 Patients Treated With a Basal-bolus Insulin Regimen
Acronym: TELESAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Sylvia Franc, Dr Sylvia Franc, MD, VP, scientific affairs, Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCOMPL06211
Record Dates: First submitted 2014-11-06; First posted 2014-11-10 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- DIABEO software alone (Experimental): Patient will have an introductory training session in the use of DIABEO by the investigating physician an will return for an on site consultation at 6 mounths (optional), 12 mounths and 24 mounths
  Interventions: Device: DIABEO software
- DIABEO+paramedical telemonitoring (Experimental): Patient will have an on site introductory training session in the use of DIABEO, by his/her "telemedicine" nurse from his/her region. The nurse will then follow up the patient according to a delegated tasks protocol written by the investigating physician with the nurse. Patient will be asked to return to see the investigator at 6 mounths (optional), 12 mounths and 24 mounths
  Interventions: Device: DIABEO software
- Usual Follow up (No Intervention): Patient will continue his/her usual follow up and return to see the investigator at 6 mounths (optional) and at the one year end of follow up for the study

INTERVENTIONS:
Device: DIABEO software — DIABEO is an electronic diary system incorporating an immediate automatic aid to calculating the insulin dose according to the prescription given by the doctor, and a data processing, automated analysis message and secure internet data transfer system. DIABEO software could be combined with remote paramedical monitoring of data (telemonitoring)
  Arms: DIABEO software alone; DIABEO+paramedical telemonitoring

SUMMARY:
The aim of the TELESAGE study is to demonstrate

1. the superiority of follow up with the DIABEO system (software alone) versus usual follow up in terms of improvement in HbA1c after 1 year in DM1 or DM2 patients treated with a basal-bolus insulin regimen.
2. the superiority of follow up with the DIABEO system (software + telemonitoring) compared to usual follow up in terms of improvement in HbA1c after 1 year in DM1 or DM2 patients treated with a basal-bolus insulin regimen.

The DIABEO software alone is an electronic diary system incorporating an immediate automatic aid to calculating the insulin dose according to the prescription given by the doctor, and a data processing, automated analysis message and secure internet data transfer system.

The DIABEO software added by paramedical telemonitoring is the electronic diary combined with remote paramedical monitoring of data (telemeonitoring)

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetic patients
* Performing auto-glycaemic control (at least 2 glycemias a day)
* Treated with insulin by a basal-bolus regimen for at least 1 year and using the same method of administration for at least 3 months (insulin pen or pump)
* Who have an Apple® or Androïde® Smartphone compatible, or intend to acquire one before their participation in the study
* Whose HbA1c dating of less 1 month and more than 3 months is ≥ 8%
* Who are able to understand and follow the study protocol
* Who have given their signed consent to take part in the study
* Subject affiliated to the French National Health Insurance funds or benefiting from such insurance

Exclusion Criteria:

* Age < 18 years old
* Patients who have used the DIABEO system within 6 months before inclusion
* Participation in a clinical study within 6 months, except for the Meos (or télédiab 3) study after a participation period of 6 months
* Patients who are pregnant or who wish to become pregnant during the study.
* Patients treated with human insulin A patient pre-screening register will be set up in each centre to establish the reasons for DM1/DM2 patients treated with a basal-bolus insulin regimen who are not taking part in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2013-02; Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
Efficacy data: change in HbA1c, measured at 1 year minus the value baseline | one year

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia FRANC, MD, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (107):
- France (107):
  - Centre hospitalier du Pays d'Aix, Aix-en-Provence
  - Clinique Claude Bernard, Albi
  - CHI d'Alencon, Alençon
  - Centre hospitalier d'Ales, Alès
  - Hotel Dieu, Angers
  - Cabinet médical, Antibes
  - Cabinet medical, Argentan
  - Clinique D'Argonay, Argonay
  - Centre hospitalier Henri Duffaut, Avignon
  - Centre hospitalier Louis Pasteur, Bagnols
  - CH Jeanne d'Arc, Bar-le-Duc
  - CH de Bayeux, Bayeux
  - Centre Hospitalier de la Cote Basque, Bayonne
  - Res Elgade, Bayonne
  - CHU de Besancon - Hopital Jean Minjoz, Besançon
  - Centre hospitalier de Bethune, Béthune
  - Centre hospitalier de Beziers, Béziers
  - Cabinet médical, Bordeaux
  - Cabinet médical, Boulogne/Mer
  - Clinique Pasteur, Brest
  - Cabinet medical, Caen
  - Hopital de la Cote de Nacre, Caen
  - centre Hospitalier Jean Rougier, Cahors
  - Centre hospitalier de Chalon sur Saone, Chalon-sur-Saône
  - CH de Chambery, Chambéry
  - CH Louis Pasteur, Cherbourg Octeville
  - Cabinet médical, Colmar
  - Cabinet médical, Colomiers
  - Hopital CHAL, Contamine-sur-Arve
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Centre Hospitalier de Dax, Dax
  - Cabinet médical, Dijon
  - Hopital du Bocage, Dijon
  - Centre hospitalier Louis Pasteur, Dole
  - Centre hospitalier de Douai, Douai
  - Centre hospitalier Simone Veil, Eaubonne
  - Centre Hospitalier Sud Essonne Etampes, Étampes
  - CHU de Fort-de-France, Fort-de-France
  - CH de Avranches Granville, Granville
  - Cabinet médical, Grenoble
  - CH Dptal Les Oudairies, La Roche-sur-Yon
  - CH Saint Louis, La Rochelle
  - Cabinet médical, La Teste-de-Buch
  - CHU de Grenoble - Hopital A Michallon, La Tronche
  - Centre Hospitalier du Creusot, Le Creusot
  - CH Le Mans, Le Mans
  - Cabinet médical, Lille
  - Hopital Claude Huriez, Lille
  - Centre hospitalier Lons-le-Saunier, Lons-le-Saunier
  - CHG Luneville, Lunéville
  - Clinique BOUCHARD, Marseille
  - Cabinet médical, Marseille
  - Cabinet La Bastide Verte, Marseille
  - Hopital Nord, Marseille
  - Hopital Sainte Marguerite, Marseille
  - Fondation Hopital Saint Joseph, Marseille
  - Hopital de La Timone, Marseille
  - Centre hospitalier de Meaux, Meaux
  - Hopitaux privés de Metz, Metz
  - Cabinet medical, Mérignac
  - Cabinet médical, Mérignac
  - Centre médical, Montpellier
  - Cabinet médical d'Alco, Montpellier
  - Hopital Lapeyronie, Montpellier
  - hôpital Emile Muller, Mulhouse
  - Cabinet médical, Muret
  - Cabinet médical, Nancy
  - Hopital Laennec - Saint Herblain, Nantes
  - Cabinet médical, Nantes
  - Cabinet médical, Nevers
  - CHAN Pierre Bérégovoy, Nevers
  - Hopital de l'Archet, Nice
  - Cabinet médical, Nice
  - Hopital Caremeau, Nîmes
  - Cabinet medical, Nîmes
  - Cabinet médical, Noisy-le-Grand
  - Cabinet médical, Orsay
  - Hopital Saint Louis, Paris
  - Cabinet médical, Paris
  - Centre hospitalier Pitié Salpetriere, Paris
  - Hopital Bichat Claude Berbard, Paris
  - Centre Hospitalier Francois Mitterrand, Pau
  - Hopital Saint Jean, Perpignan
  - Hôpital Haut Lévêque, Pessac
  - Hôpital Saint André, Pessac
  - Centre Hospitalier de Périgueux, Périgueux
  - Centre médical des spécialistes, Plan-de-Cuques
  - CHRA, Pringy
  - Centre hospitalier de Rambouillet, Rambouillet
  - Hopital Robert Debré, Reims
  - Hopital Sud Anne de Bretagne, Rennes
  - Hopital Victor Provo, Roubaix
  - Groupe médical ELGAR, Saint-Jean-de-Luz
  - CHU de Saint Etienne - Hopital Nord, Saint-Priest-en-Jarez
  - Cabinet de groupe, Strasbourg
  - Hôpital Civil, Strasbourg
  - Centre hospitalier de Bigorre site La Gespe, Tarbes
  - Hopital Beauregard, Thionville
  - CHITS Hopital Sainte Musse, Toulon
  - Hopital Rangueil, Toulouse
  - Hopital Joseph Ducuing, Toulouse
  - Cabinet médical, Toulouse
  - Clinique Ambroise Paré, Toulouse
  - CH de Valence, Valence
  - Centre hospitalier de Valenciennes, Valenciennes
  - Hopitaux de Brabois, Vandœuvre-lès-Nancy
  - Cabinet medical, Vénissieux

REFERENCES:
- [Derived] Jeandidier N, Chaillous L, Franc S, Benhamou PY, Schaepelynck P, Hanaire H, Catargi B, Farret A, Fontaine P, Guerci B, Reznik Y, Penfornis A, Borot S, Serusclat P, Kherbachi Y, D'Orsay G, Detournay B, Simon P, Charpentier G. DIABEO App Software and Telemedicine Versus Usual Follow-Up in the Treatment of Diabetic Patients: Protocol for the TELESAGE Randomized Controlled Trial. JMIR Res Protoc. 2018 Apr 19;7(4):e66. doi: 10.2196/resprot.9154. PMID 29674306